CLINICAL TRIAL: NCT07263360
Title: A Single-arm, Single-center Clinical Study of Iparomlimab and Tuvonralimab Injection Combined With GemOX and Lenvatinib as Conversion Therapy for Initially Potentially Resectable Intrahepatic Cholangiocarcinoma and Gallbladder Cancer
Brief Title: Iparomlimab and Tuvonralimab Injection Combined With GemOX and Lenvatinib as Conversion Therapy for Initially Potentially Resectable Intrahepatic Cholangiocarcinoma and Gallbladder Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20251152
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: BTC
Keywords: lparomlimab and Tuvonralimab injection; GemOX; Lenvatinib
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab Injection combined with GemOX and lenvatinib (Experimental): Iparomlimab and Tuvonralimab Injection combined with GemOX and lenvatinib
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection combined with GemOX and lenvatinib

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection combined with GemOX and lenvatinib — Iparomlimab and Tuvonralimab Injection:5 mg/kg, intravenous infusion on Day 1 of each 3-week cycle (q3w); for 4 to 6 cycles.
  Lenvatinib: 8-12 mg, orally once daily (qd). The dose is determined by body weight:8 mg po qd for body weight < 60 kg;12 mg po qd for body weight ≥ 60 kg
  GemOX Regimen:
  Oxaliplatin: 85 mg/m², intravenous infusion on Day 1 of each 3-week cycle (q3w); for a maximum of 6 cycles.
  Gemcitabine: 1000 mg/m², intravenous infusion on Day 1 and Day 8 of each 3-week cycle (q3w); for a maximum of 6 cycles.
  Postoperative Treatment for Patients with Successful Conversion:
  Iparomlimab and Tuvonralimab Injection: 5 mg/kg, intravenous infusion on Day 1 of each 3-week cycle (q3w); for 8 cycles.
  For Patients without Successful Conversion:
  Subsequent treatment regimens will be determined by the investigator.

SUMMARY:
The primary objective is to evaluate the efficacy and safety of Iparomlimab and Tuvonralimab Injection (QL1706, an Anti-PD-1/CTLA-4 Combined Antibody) combined with GemOX and lenvatinib as conversion therapy for Initially Potentially Resectable intrahepatic cholangiocarcinoma and gallbladder cancer.

DETAILED DESCRIPTION:
This single-arm, single-center clinical study aims toevaluate the efficacy and safety of Iparomlimab and Tuvonralimab Injection (QL1706, an Anti-PD-1/CTLA-4 Combined Antibody) combined with GemOX and lenvatinib as conversion therapy for Initially Potentially Resectable intrahepatic cholangiocarcinoma and gallbladder cancer. This study consists of three phases: screening, treatment, and follow-upEfficacy evaluation and safety monitoring should be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, male or female.
* Histologically or cytologically confirmed diagnosis of locally advanced or potentially resectable intrahepatic cholangiocarcinoma or gallbladder cancer, defined as T2b-T4 or N1 M0 according to the AJCC 8th edition.
* Expected life expectancy ≥ 12 weeks.
* No prior systemic treatment for biliary tract cancer before the first dose of study medication.
* At least one measurable lesion as defined by RECIST 1.1 criteria.
* ECOG Performance Status of 0 or 1.
* Adequate organ function, without severe dysfunction of the hematologic, cardiac, pulmonary, hepatic, renal, bone marrow, or immune systems.
* Laboratory tests meeting the following requirements: Women of childbearing potential must have a negative pregnancy test (serum or urine) within 14 days before enrollment and voluntarily use adequate contraception during the observation period and for 8 weeks after the last dose of the study drug. For men, they must be surgically sterile or agree to use adequate contraception during the observation period and for 8 weeks after the last dose of the study drug.
* Patient voluntarily participates and provides written informed consent.
* Good compliance is anticipated, allowing for efficacy and adverse event follow-up per the protocol.

Exclusion Criteria:

* The subject has received any prior antitumor therapy or any investigational anticancer agents.
* Presence of any active autoimmune disease or a history of autoimmune diseases (e.g., interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism [may be enrolled if stable on hormone replacement therapy]). Patients with childhood asthma that has completely resolved in adulthood without any intervention, or vitiligo, may be enrolled. Patients requiring medical intervention with bronchodilators are not eligible.
* Known congenital or acquired immunodeficiency, such as Human Immunodeficiency Virus (HIV) infection.
* Uncontrolled cardiac clinical symptoms or diseases, e.g., NYHA Class II or above heart failure, unstable angina, myocardial infarction within 1 year, or patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention.
* Severe concurrent infection within 4 weeks prior to the first dose (e.g., requiring intravenous antibiotics, antifungals, or antivirals), or unexplained fever >38.5°C during screening/prior to the first dose.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Administration of a live attenuated vaccine within 4 weeks prior to the first dose or planned administration during the study period.
* History of or concurrent other malignant tumors within the past 5 years (except for adequately treated basal cell carcinoma of the skin, carcinoma in situ of the cervix, and ovarian cancer).
* Gastrointestinal bleeding event or active hemoptysis within 28 days prior to the first dose.
* Gastric or esophageal varices requiring treatment.
* Active malignant tumors within 36 months prior to enrollment.
* Known allergy to any of the investigational drug components.
* Poorly controlled psychiatric disorder.
* Presence of superior mesenteric vein tumor thrombus, metastasis to group 16 lymph nodes, or distant metastasis to other organs / biological factors: peritoneal metastasis, direct invasion to adjacent organs, etc. / involvement of organs (pancreas, stomach, duodenum, colon) that cannot be resected en bloc.
* Any other condition deemed by the investigator as unsuitable for enrollment. This includes, but is not limited to, pre-existing central nervous system metastases, severe laboratory abnormalities, or familial/social factors that could compromise the subject's safety, or data/sample collection.
* Patients with extensive liver metastases involving the entire liver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate | up to 12 month

SECONDARY OUTCOMES:
Conversion Rate | up to 12 month
Objective response rate | up to 12 month
  the percentage of participants in the analysis population who had a CR(Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) usingRECIST 1.1 based on investigator assessment.
Progression-Free Survival | up to 12 month
  PFS was defined as the time from first dose of study treatment to the firstdocumented PD per REClST 1.1 by investigator assessment, or death due to any cause, whicheveroccurred first.
pathological Complete Response | up to 12 month
Overall survival | up to 36 month
  OS was defined as the time from the first dose of study drug to death due to any cause.
Adverse Events | up to 36 month
  An AE was defined as any untoward medical occurrence in a pharmaceutical productwhich does not necessarily have to have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No